CLINICAL TRIAL: NCT05131464
Title: An Open-label, Single-arm, Multicenter, Extension Study to Evaluate the Long-term Safety and Efficacy of CM310 in Patients With Chronic Rhinosinusitis With Nasal Polyps
Brief Title: The Study of CM310 in Patients With Chronic Rhinosinusitis With Nasal Polyps
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM310NP100
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2023-12

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM310 (Experimental)
  Interventions: Drug: CM310

INTERVENTIONS:
Drug: CM310 — CM310, 300 mg/2 mL, SC, every 2 weeks

SUMMARY:
This is an open-label, single-arm, multicenter, extension study to evaluate the long-term safety and efficacy of CM310 in patients with CRSwNP.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be able to understand and voluntarily sign an ICF.
* Participated in the clinical study of CM310 in patients with CRSwNP (Study No. of CM310NP001) and meet the criterion "a" or "b" as below:

  1. Patients have completed the treatment as required by the protocol and completed the EOS (V12) visit;
  2. Early withdrawal from the visit due to poor compliance or other objective reasons other than CM310-related AE, and the patient have completed early withdraw visit as per protocol, and, as assessed by the investigator and sponsor, the factors resulting in early termination of main study treatment have disappeared/will not affect the patient's participation in this extension study.
* Patients must have received INCS at a relatively stable dose for at least 4 weeks upon the screening visit.

Exclusion Criteria:

* Patients who are considered ineligible for continuous CM310 treatment by the investigator and the sponsor due to CM310-related* SAE or discontinuation caused by CM310-related* AE developed in the main study.
* Patients who had poor compliance in the main study and are judged unable to complete this study by the investigator.
* Not enough washing-out period for previous therapy.
* Presence of other concomitant and poorly controlled serious diseases or recurrent chronic diseases, including but not limited to active infections, cardiovascular and cerebrovascular diseases, pulmonary tuberculosis or other pathogen infections, diabetes mellitus, autoimmune diseases, human immunodeficiency virus (HIV) infection, active hepatitis B, hepatitis C or parasitosis, neoplasm malignant, etc.
* Patients with severe hepatic or renal impairment, characterized by aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level > 2 times of upper limit of normal (ULN) or serum creatinine level > ULN.
* Women who are pregnant or breastfeeding, or who plan to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Incidences of TEAE, SAE and AESI related to CM310; Abnormalities in laboratory tests, physical examination, vital sign and 12-lead electrocardiogram. | approximately 2 years
  Incidences of TEAE, SAE and AESI related to CM310; Abnormalities in laboratory tests, physical examination, vital sign and 12-lead electrocardiogram.

SECONDARY OUTCOMES:
Changes from baseline in total nasal polyp score (NPS) from both sides at each evaluation time point. | approximately 2 years
  The NPS score will be graded based on the nasal polyp size of both left and right nostrils described by nasal endoscopy by the study doctor nasal endoscopy. Each nostril is scored on a scale of 0-4, with the total score being the sum of both nostrils (0-8).
Changes from baseline in weekly average nasal congestion score (NCS) at each evaluation time point. | approximately 2 years
  The NCS scoring ranges from 0-3 points and is conducted separately on both left and right nostril. The higher score from either left or right side is taken as the NCS score on each day, and the total score is 3 points.
Changes from baseline in University of Pennsylvania Smell Identification Test (UPSIT) score at each evaluation time point. | approximately 2 years
  The UPSIT has a total of 40 questions and consists of 4 different booklets. The test patient will smell the odorant level after cutting the capsule with a nail or pencil and then choose an answer from 4 choices on each page. One score is counted if an odor is correctly selected, with a total score of 40 points. The lower the score, the more impaired the smell function.
Changes from baseline in sino-nasal outcome test-22 (SNOT-22) score at each evaluation time point. | approximately 2 years
  The SNOT-22 score is a specific scale for chronic rhinosinusitis and can evaluate the patient-reported outcome (PRO) and health-related quality of life (HRQoL) of patients suffering from chronic rhinosinusitis, with contents covering 22 dimensions related to quality of life. Each dimension is scored as 0-5, so with a total score of 110.
Changes from baseline in patient's nasal total symptom score (TSS) at each evaluation timepoint. | approximately 2 years
  The evaluation content of TSS includes three aspects: nasal congestion, loss of smell and running nose. Each aspect has a score of 0-3 with a total score of 0-9. The higher score indicates the more severe overall symptom.
Changes from baseline in Lund-Mackay score of sinus CT scan at each evaluation time point. | approximately 2 years
  Sinus CT scan evaluation includes Lund-Mackay scores and 3D volumetric measurement of the sinus, which are objective evaluation parameters commonly used to evaluate the severity of CRS.
Changes from baseline in three-dimensional sinus inflammation volume of sinus CT scan performed sat each evaluation time point. | approximately 2 years
  Sinus CT scan evaluation includes Lund-Mackay scores and 3D volumetric measurement of the sinus, which are objective evaluation parameters commonly used to evaluate the severity of CRS.
Changes from baseline in total scores of NPS and NCS in patients with a nasal polyp surgery history or complication with asthma at each evaluation time point. | approximately 2 years
Percentage of patients receiving rescue therapy. | approximately 2 years
Immunogenicity endpoint: generation of anti-drug antibodies (ADAs) and/or neutralizing antibodies (Nabs). | approximately 2 years
PD endpoint: Changes from baseline in eosinophils levels in plasma and nasal polyp biopsy samples at each evaluation time point. | approximately 2 years
PK endpoint: steady-state trough concentration (CtroughSS) of CM310. | approximately 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Tong-Ren hospital, Beijing
  - Site 3, Chengdu
  - Site 2, Wuhan